CLINICAL TRIAL: NCT05740319
Title: Efficacy and Safety Evaluation of Fecal Microbiota Transplantation in Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-507R
Record Dates: First submitted 2023-02-09; First posted 2023-02-23 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT (Experimental): Participants will be given FMT through oral capsules or nasojejunal tube once a month for three months.
  Interventions: Other: FMT

INTERVENTIONS:
Other: FMT — FMT refers to transplanting healthy donor-derived microbiota to participants via oral capsule or injection of fecal suspension via nasojejunal tube.

SUMMARY:
Participants will be given FMT through oral capsules or nasojejunal tube once a month. After three-time treatment, participants were followed up for three months. Participants complete specific scales to assess improvement in symptoms, emotion and quality of life. Besides, they report adverse effects and collect fecal samples at each visit.

DETAILED DESCRIPTION:
This prospective, single-arm interventional study aims to evaluate efficacy and safety of fecal microbiota transplantation in refractory IBS patients. Patients meeting the inclusion and exclusion criteria will provide written informed consent and receive FMT from healthy donors for three times. The administration methods include taking oral capsule or delivering microbiota suspension into the duodenum via nasojejunal tube. The patients receive treatment once a month and will be followed up for 3 months. Improvement in IBS symptoms, emotion and quality of life were assessed through IBS symptom severity scale (IBS-SSS), Gastrointestinal symptom rating scale (GSRS), IBS-Global Assessment of Improvement (IBS-GAI), Self-rating Anxiety Scale (SAS), Self-rating Depression Scale (SDS) and IBS-Quality of Life (IBS-QoL) respectively. Patients were asked to complete these scales and collect fecal samples at baseline, post-FMT and at 1, 2, 3 and 4 months after FMT. Primary endpoints were improvement in IBS-SSS score and global symptoms after three-time FMT. Secondary endpoints include Change in GSRS score, improvement in emotion and quality of life at post-FMT, 1 and 6 months, as well as change in fecal microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfilled the Rome IV criteria for the diagnosis of IBS, aged 18-70 years;
* Patients who have experienced failure of at least 3 conventional therapies for IBS;
* Absence of red flags such as weight loss, hematochezia;

Exclusion Criteria:

* Pregnant, planning pregnancy or lactating;
* Psychiatric disorder or unable to cooperate with treatment and follow-up visit;
* Immunodeficiency or treatment with immune-modulating medication;
* Use of probiotics within the previous 3 months or treatment with antibiotics within 1 month prior to study entry;
* Having undergone any abdominal surgery, with the exception of appendectomy, cholecystectomy, caesarean section and hysterectomy;
* Presence of uncontrolled diabetes, hypertension, thyroid disease or other systemic disease;
* Presence of severe diseases related to heart, brain, kidney and lung or concomitant malignancies;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline IBS symptom severity scale (IBS-SSS) score at 9 weeks | at baseline and 9 weeks
  IBS symptom severity scale (IBS-SSS) is used to evaluate change in IBS symptoms, with a score ranging from 0 to 500. Higher score means severer IBS symptom. Change in IBS-SSS score is obtained by evaluating the scale at baseline and 9 weeks (after three-time FMT).
Response rate at 9 weeks | at 9 weeks
  Investigator ask participants a single question, "Compared to the way you felt before you entered the study, have you IBS symptoms over the past 7 days been: 1)"Substantially Worse"; 2)"Moderately Worse"; 3) Slightly Worse; 4)"No Change"; 5) Slightly Improved"; 6) Moderately Improved"; 7) Substantially Improved". Responder is defined as participants who report "moderately improved" or "substantially improved".

SECONDARY OUTCOMES:
Change from baseline IBS symptom severity scale (IBS-SSS) score at 1 week, 1 month and 6 months | at baseline, 1 week, 1 month and 6 months
  IBS symptom severity scale (IBS-SSS) is used to evaluate change in IBS symptoms, with a score ranging from 0 to 500. Higher score means severer IBS symptom. Change in IBS-SSS score is obtained by evaluating the scale at baseline and at 1 week (after first FMT), 1 month (three weeks after first FMT), and 6 months (4 months after three-time FMT).
Change from baseline Gastrointestinal Symptom Rating Scale (GSRS) score at 1 week, 1 month, 9 weeks and 6 months | at baseline, 1 week, 1 month, 9 weeks and 6 months
  Gastrointestinal symptom rating scale (GSRS) is used to evaluate change in gastrointestinal symptoms, with a score ranging from 15 to 105. Higher score means severer gastrointestinal symptoms. Change in IBS-SSS score is obtained by evaluating the scale at baseline, 1 week (after first FMT), 1 month (three weeks after first FMT), 9 weeks (after three-time FMT) and 6 months (4 months after three-time FMT).
Change from baseline IBS-Quality of Life (IBS-QoL) score at 1 month, 3 months and 6 months | at baseline, 1 month, 3months and 6 months
  IBS-Quality of Life (IBS-QoL) is a specific scale used to evaluate change in quality of life, with a score ranging from 0 to 100. Higher score indicates worse quality of life. Change in IBS-QoL score is obtained by evaluating the scale at baseline, 1 month (three weeks after first FMT), 3 months (three weeks after third FMT) and 6 months (4 months after three-time FMT). An over-14-point reduction is considered a significant improvement in quality of life.
Change from baseline Self-rating Anxiety Scale (SAS) score at 1 month, 3 months and 6 months | at baseline, 1 month, 3months and 6 months
  Self-rating Anxiety Scale (SAS) is used to evaluate change in IBS-related anxiety, with a score ranging from 25 to 100. Higher score indicates higher level of anxiety. Change in SAS score is obtained by evaluating the scale at baseline, 1 month (three weeks after first FMT), 3 months (three weeks after third FMT) and 6 months (4 months after three-time FMT).
Change from baseline Self-rating Depression Scale (SDS) score at 1 month, 3 months and 6 months | at baseline, 1 month, 3months and 6 months
  Self-rating Depression Scale (SDS) is used to evaluate change in IBS-related depression, with a score ranging from 25 to 100. Higher score indicates higher level of depression. Change in SDS score is obtained by evaluating the scale at baseline, 1 month (three weeks after first FMT), 3 months (three weeks after third FMT) and 6 months (4 months after three-time FMT).
Response rate at 1 week, 1month, 3 months and 6 months | at 1 week, 1month, 3 months and 6 months
  Investigator ask participants a single question, "Compared to the way you felt before you entered the study, have you IBS symptoms over the past 7 days been: 1)"Substantially Worse"; 2)"Moderately Worse"; 3) Slightly Worse; 4)"No Change"; 5) Slightly Improved"; 6) Moderately Improved"; 7) Substantially Improved". Responder is defined as participants who report "moderately improved" or "substantially improved".
Change from baseline fecal microbiota composition at 1 week, 1 month and 6 months | at baseline, 1 week, 1 month and 6 months
  Fecal samples are collected at baseline, 1 week (after first FMT), 1 month (three weeks after first FMT) and 6 months (4 months after three-time FMT). Change in fecal microbiota was measured by 16S rRNA sequencing and metagenomics.
Change from baseline fecal metabolites at 1 week, 1 month and 6 months | at baseline, 1 week, 1 month and 6 months
  Fecal samples are collected at baseline, 1 week (after first FMT), 1 month (three weeks after first FMT) and 6 months (4 months after three-time FMT). Change in fecal metabolites are measured by untargeted metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Dong, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No